CLINICAL TRIAL: NCT03941145
Title: Effectiveness of a Novel Workplace-based Exercise Intervention: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Stirling (Other)
Collaborators: Swansea University (Other)
Responsible Party: Principal Investigator, Niels Vollaard, Principal Investigator, University of Stirling
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18/19 036
Record Dates: First submitted 2019-04-26; First posted 2019-05-07 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Health Behavior
Keywords: exercise
MeSH Terms: conditions — Health Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Participants allocated to the intervention group will be asked to perform 2 exercise sessions per week for 6 weeks. Each session will involve 10 min of low-intensity cycling (25 W) interspersed with two 20-s 'all-out' cycle sprints against a resistance equivalent to 5% of body mass. The exercise intervention will be delivered on a commercially available cycle ergometer with software developed by CAR.O.L.
  Interventions: Behavioral: Reduced-Exertion High-Intensity Interval Training (REHIT)
- Control (No Intervention): The effects of the intervention will be compared to a no-intervention control group recruited from the same workplace settings.

INTERVENTIONS:
Behavioral: Reduced-Exertion High-Intensity Interval Training (REHIT) — REHIT is a type of Sprint Interval Training (SIT) that has been shown to be efficacious at improving maximal aerobic capacity using a minimal volume of exercise.
  Arms: Exercise

SUMMARY:
Sufficient physical activity and a good cardiorespiratory fitness level (CRF) are central in cardiovascular disease (CVD) risk reduction. However, many people remain inactive, partly because current exercise recommendations fail to address important barriers to exercise. A novel exercise protocol has previously been developed called 'reduced-exertion high-intensity interval training' (REHIT), which can remove several common perceived barriers to exercise. REHIT 1) improves CRF and other key CVD risk factors, 2) is genuinely time-efficient (total time-commitment of just 2x10 min per week), 3) is well-tolerated, manageable, and not associated with negative affective responses, and 4) can be done in the workplace, in work-clothes and without a need to shower afterwards. To date, this intervention has only been investigated in a lab-setting. Therefore, in the present randomised controlled trial, the 'real-world' effectiveness of REHIT in improving maximal aerobic capacity (V̇O2max; a key risk factors of CVD) will be investigated in a workplace setting. Participants' attitudes and psychological responses to REHIT will be assessed to evaluate the likelihood of successful implementation. In 2 study centres, a total of up to n=50 physically inactive male and female office workers will be recruited to perform 6 weeks of unsupervised, computer-guided, office-based REHIT (n=25) or act as a control (n=25).

ELIGIBILITY:
Inclusion Criteria:

• Employee at participating workplace

Exclusion Criteria:

* Aged < 18 years or > 60 years
* History of type 2 diabetes
* Insulin therapy
* Use of β-blockers
* Use of inhaled steroids (e.g. for asthma)
* Any cardiovascular condition with the exception of well-controlled uncomplicated hypertension (systolic >140 mm Hg and/or >90 mm Hg after at least 5 minutes of seated rest), which is treated with no more than two drugs (either an ACE, ARB, calcium channel blocker, or diuretic)
* Cerebrovascular disease including previous stroke or aneurysm
* History of exercise-induced asthma
* History of type 1 diabetes mellitus or a history of ketoacidosis
* History of other specific types of diabetes (e.g., genetic syndromes, secondary pancreatic diabetes, diabetes due to endocrinopathies, drug or chemical-induced, and post organ transplant)
* History of respiratory disease including pulmonary hypertension or chronic obstructive pulmonary disease
* History of musculoskeletal or neurological disorders
* Active inflammatory bowel disease
* History of renal disease
* Other metabolic diseases, including hyper/ hypo-parathyroidism, hyper/hypo-thyroidism, and Cushing's disease.
* BMI>35 kg/m2
* A clinically significant resting ECG abnormality at the pre-screening visit which in the opinion of the cardiologist exposes the participant to risk by take part in the main trial.
* 'Yes' to any questions on a standard physical activity readiness questionnaire (PARQ)
* Classification as moderately or highly physically active on the International Physical Activity Questionnaire (IPAQ)
* Current participation in another research study
* Inability to fully understand the verbal and written descriptions of the study in English, and the instructions provided during the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-09-13 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
Change in maximal aerobic capacity | Change from baseline to 3 days after the 6-week intervention
  Aerobic capacity: a key risk factor of noncommunicable disease

SECONDARY OUTCOMES:
Change in motivation for exercise | Change from baseline to 3 days after the 6-week intervention
  Motivation to exercise as assessed using the RM 4-FM questionnaire, a 16-item questionnaire assessing reasons for trying to be physically active on a scale from 1 ('not at all true') to 7 ('very true'). Higher scores indicate a greater motivation for performing exercise. Scores are added to get an overall score, with higher overall scores indicating greater intrinsic motivation.
Change in health status | Change from baseline to 3 days after the 6-week intervention
  Health status as assessed using the Short Form (36) Health Survey (SF36), which is a 36-item, patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Change in perceived stress | Change from baseline to 3 days after the 6-week intervention
  Perceived stress as assessed using the Perceived Stress Scale questionnaire, which measures the degree to which situations in one's life are appraised as stressful. The 10-item questionnaire ask for the frequency of stressful events in the last month, scored on a scale from 0 ('never') to 4 ('very often'). The sum score is taken, with higher scores indicating more perceived stress.
Intervention acceptability | 3 days after the 6-week intervention
  Intervention acceptability as assessed using a questionnaire published by Boereboom et al (2016). This 11-item questionnaire asks how strongly participants agree with statements on the acceptability of the exercise intervention on a scale from 1 ('strongly disagree') to 5 ('strongly agree').

CONTACTS AND LOCATIONS:
Locations (1):
- Stirling Council, Stirling, United Kingdom

IPD SHARING:
Plan to Share IPD: No
data will be disseminated / published as means +- SD. no individual data will be presented.

REFERENCES:
- [Derived] Metcalfe RS, Atef H, Mackintosh K, McNarry M, Ryde G, Hill DM, Vollaard NBJ. Time-efficient and computer-guided sprint interval exercise training for improving health in the workplace: a randomised mixed-methods feasibility study in office-based employees. BMC Public Health. 2020 Mar 12;20(1):313. doi: 10.1186/s12889-020-8444-z. PMID 32164631